CLINICAL TRIAL: NCT06933056
Title: Comparison of Antiplatelet Effects of Sotagliflozin to FDA-approved Antiplatelet Drugs: an Interventional Study
Brief Title: Comparison of Antiplatelet Effects of Sotagliflozin to FDA-approved Antiplatelet Drugs
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Lexicon Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Michael Holinstat, Professor of Pharmacology, Professor of Internal Medicine and Professor of Surgery, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00267102
Record Dates: First submitted 2025-04-04; First posted 2025-04-18 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Platelet Function and Reactivity Tests
Keywords: Sotagliflozin
MeSH Terms: interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; apixaban

STUDY DESIGN:
Intervention Model Description: administration of antiplatelet and anticoagulant drugs given to subjects in randomized order with washout period between drug administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Platelet function in healthy subjects administered sotagliflozin vs. antiplatelet agents (Experimental): Platelet responsiveness will be assessed in the blood from subjects administered sotagliflozin, aspirin, clopidogrel, or apixaban in randomized order given as a single drug administration.
  Interventions: Drug: Sotagliflozin (SOTA) followed by 3 drugs in a random order; Drug: Aspirin followed by 3 drugs in a random order; Drug: Clopidogrel followed by 3 drugs in a random order; Drug: Eliquis followed by 3 drugs in a random order

INTERVENTIONS:
Drug: Sotagliflozin (SOTA) followed by 3 drugs in a random order — 400 mg/day SOTA Each drug will be given daily for 2 weeks.
Drug: Aspirin followed by 3 drugs in a random order — 81 mg/day Aspirin Each drug will be given daily for 2 weeks.
Drug: Clopidogrel followed by 3 drugs in a random order — 75 mg/day clopidogrel Each drug will be given daily for 2 weeks.
Drug: Eliquis followed by 3 drugs in a random order — 5 mg orally twice daily Eliquis Each drug will be given daily for 2 weeks.
  Other Names: Apixaban

SUMMARY:
This study will identify the potential benefits of regulating platelet activation with sotagliflozin compared to other FDA-approved drugs known to limit platelet activation.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Students under the direct supervision of Dr. Michael Holinstat
* Subjects diagnosed with Type I diabetes or those with ketoacidosis
* Subjects with a history of alcohol abuse, pancreatitis or pancreatic surgery, or subjects taking a ketogenic diet
* Women who self-identify as being pregnant or who are planning to become pregnant during the 14 week study will be excluded from the study, as are those who are breastfeeding (women enrolled in the study will be given a urine pregnancy test at the start of each drug administration period to confirm pregnancy status)
* Subjects with hypersensitivity to aspirin, clopidogrel, apixaban, or sotagliflozin are excluded
* have active bleeding, or who have who have a history of balanitis or balanoposthitis, genital mycotic infections, or a planned elective surgical/dental procedure 1 month prior to or following completion of study
* Subjects who have taken Non-Steroidal Anti-Inflammatory Drugs (NSAIDS; examples of NSAIDS are Ibuprofen (Advil, Motrin) and Naproxen (Aleve)) or aspirin within 7 days prior to the study or anticoagulants within 10 days prior to the study
* individuals currently taking SSRI's (for example, Fluoxetine (Prozac), Sertraline (Zoloft), Paroxetine (Paxil), Citalopram (Celexa), and Escitalopram (Lexapro).), SNRI's (Duloxetine (Cymbalta), Venlafaxine (Effexor XR), Desvenlafaxine (Pristiq), and Levomilnacipran (Fetzima)), lithium, or omeprazole/esomeprazole
* Subjects less than or equal to 60 kg will be excluded
* Subjects with a creatinine greater than or equal to 1.5 mg/dl will be excluded

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Platelet aggregation | Blood will be drawn and aggregation measured at baseline (day 1) and every 14 days.
  Measured from blood samples

SECONDARY OUTCOMES:
Platelet granule secretion | Blood will be drawn and granule secretion measured at baseline (day 1) and every 14 days.
  Measured from blood samples
Total thrombus activation with T-TAS | Blood will be drawn and T-TAS measured at baseline (day 1) and every 14 days.
  Measured from blood samples
Thromboelastography (TEG) | Blood will be drawn and thromboelastography measured at baseline (day 1) and every 14 days.
  Measured from blood samples
Platelet integrin activation | Blood will be drawn and platelet integrin activation measured at baseline (day 1) and every 14 days.
  Measured from blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Michael Holinstat, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No